CLINICAL TRIAL: NCT02910245
Title: Efficacy of Optimized Thiopurine Therapy in Ulcerative Colitis (OPTIC)
Brief Title: Mercaptopurine Therapy in Ulcerative Colitis
Acronym: OPTIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, M. Lowenberg, Gastroenterologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SA652012
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Colitis, Ulcerative
Keywords: Therapeutic Drug Monitoring; Mercaptopurine (6-MP); Thiopurine; Efficacy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mercaptopurine; Mesalamine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mercaptopurine (Purinethol) (Active Comparator): Mercaptopurine (Purinethol),1-1.5 mg/kg/day oral, 52 weeks & Prednisone, 40 mg/day oral, 2 weeks, followed by fixed tapering over 6 weeks OR budesonide (cortiment) 9 mg/day during 8 weeks & Mesalamine, 2 g/day oral, 52 weeks.
  Interventions: Drug: Mercaptopurine (Purinethol); Drug: Mesalamine; Drug: Prednisone
- Placebo (Placebo Comparator): Placebo, 1-1.5 mg/kg/day, 52 weeks & Prednisone, 40 mg/day oral, 2 weeks, followed by fixed tapering over 6 weeks OR budesonide (cortiment) 9 mg/day during 8 weeks & Mesalamine, 2 g/day oral, 52 weeks.
  Interventions: Drug: Placebo; Drug: Mesalamine; Drug: Prednisone

INTERVENTIONS:
Drug: Mercaptopurine (Purinethol)
  Other Names: Purinethol
  Arms: Mercaptopurine (Purinethol)
Drug: Placebo
  Arms: Placebo
Drug: Mesalamine
  Other Names: Asacol; Mezavant; Pentasa; Salofalk
Drug: Prednisone

SUMMARY:
This project is a double-blind, randomized, placebo-controlled, multicenter trial in the Netherlands. The aim of this study is to investigate the therapeutic efficacy of optimized 6-mercaptopurine (6-MP) in ulcerative colitis patients. Therapeutic drug monitoring (TDM) will be performed in order to optimize treatment outcomes and objective endoscopic endpoints will be used.

DETAILED DESCRIPTION:
Subjects will receive treatment with oral prednisone 40 mg/day for 2 weeks, followed by fixed tapering over 6 weeks. Half of the subjects will be randomized to concomitant 6-MP 1-1.5 mg/kg/day and half will receive concomitant placebo treatment. During the entire course of the trial all subjects will receive maintenance treatment with 5-ASA in an oral dose of at least 2 gram per day. Subjects will be subjected to one colonoscopy at baseline and one sigmoidoscopy in week 52 in order to assess endoscopic disease activity.

Data will be collected using electronic case report forms (eCRF) with Castor EDC. Quality and data validation procedures will be applied to ensure the validity and accuracy of the clinical database. Monitoring of the study will be done according to the GCP guidelines and following a monitoring plan. The financier of the study, ZonMw Goed Gebruik Geneesmiddelen, has the right to perform an audit if seen necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of UC by endoscopy and histopathology
2. Patients between 18 and 80 years of age
3. Active disease, despite oral treatment with at least 2g/day 5-ASA
4. Treatment with oral corticosteroids is required

Exclusion Criteria:

1. Prior treatment with thiopurines
2. Prior treatment with biologics (e.g. anti-TNF agents and vedolizumab)
3. Current pregnancy (a pregnancy test will be performed if necessary according to the treating physician)
4. Chronic Obstructive Pulmonary Disease (COPD)
5. Acute coronary heart disease
6. (Bacterial) gastroenteritis has to be treated first
7. Coagulation disorders
8. Active malignancy
9. History of colonic dysplasia/cancer
10. Extensive colonic resection, i.e. subtotal colectomy with <15 cm colon in situ
11. Concomitant therapy with drugs interfering with MP metabolism, like allopurinol, ribavirin or anti-epileptics.
12. Known systemic fungal infections or parasitic infections have to be treated first
13. Known duodenal or ventricular ulcus
14. Substance abuse, such as alcohol (> 80 gram/day - one standard glass contains 10 gram of alcohol), I.V. drugs and inhaled drugs. If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 2 years. Subjects receiving methadone within the past 2 years are also excluded
15. Positive tuberculosis screen (when a screening is performed at the discretion of the treating physician)
16. Active hepatitis B virus or hepatitis C virus infection defined as a positive anti-HCV, HBsAg and/or anti-HBcore screening.
17. Leucopenia (Neutrophil count < 1,8x10^9/L)
18. Thrombopenia (Platelets < 90x10^9/L)
19. Elevated liver enzymes (>2x ULN)
20. Abnormal renal function (eGFR< 30 mL/min)
21. Other conditions which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical and endoscopic remission | After 52 weeks of treatment
  Defined as a SCCAI-score ≤ 4, a UCEIS-score ≤ 3 and a total Mayo score ≤ 2, with no individual subscore >1.

SECONDARY OUTCOMES:
(Serious) Adverse Events | Continue during 52 weeks of treatment
  Occurrence of (serious) adverse events ((S)AE)
Leukocyte counts | Every 6 weeks during 52 weeks of treatment
Liver function tests | Every 6-12 weeks during 52 weeks of treatment
Occurrence of subjective thiopurine intolerance | Every 6-12 weeks during 52 weeks of treatment
6-TGN levels | Every 6-12 weeks during 52 weeks of treatment
6-MMP levels | Every 6-12 weeks during 52 weeks of treatment
Occurrence of treatment failure | Continue during 52 weeks of treatment
Occurrence of upscaling treatment | Continue during 52 weeks of treatment
  Occurrence of upscaling treatment to biologicals (anti-TNF agents or vedolizumab)
Treatment costs | Every 3 months during 52 weeks of treatment
  Budget-impact analysis and cost-utility analysis

OTHER OUTCOMES:
Disease specific quality of life | Every 3 months during 52 weeks of treatment
  Quality of life measured by use of the IBD questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Löwenberg, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (12):
- Netherlands (12):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander MC, Amersfoort
  - Amsterdam UMC, location VUMC, Amsterdam
  - OLVG Oost, Amsterdam
  - Amsterdam UMC, location AMC, Amsterdam
  - Amstelland Hospital, Amsterdam
  - Tergooi Hospital, Hilversum
  - Westfriesgasthuis, Hoorn
  - St. Antonius Hospital, Nieuwegein
  - Sint Franciscus Gasthuis, Rotterdam
  - MC Haaglanden, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523